CLINICAL TRIAL: NCT01534143
Title: A Pilot Study Using High Dose Busulfan and Bortezomib as Part of Allogeneic Transplant Conditioning Regimen for High Risk Multiple Myeloma Patients.
Brief Title: High Dose Busulfan and Bortezomib in Treating Patients With High Risk Multiple Myeloma Undergoing Stem Cell Transplant
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Data was not collected, because funding was unavailable to continue study.
Sponsor: Barbara Ann Karmanos Cancer Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Zaid Al-Kadhimi, Principal Investigator, Barbara Ann Karmanos Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2011-151; NCI-2012-00120 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2012-02-13; First posted 2012-02-16 (Estimated); Results first posted 2013-12-16 (Estimated); Last update posted 2017-04-05 (Actual); Status verified 2017-03

CONDITIONS: Refractory Multiple Myeloma; Stage I Multiple Myeloma; Stage II Multiple Myeloma; Stage III Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — Tacrolimus; Sirolimus; Antilymphocyte Serum; thymoglobulin; fludarabine phosphate; Busulfan; Bortezomib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (chemotherapy, enzyme inhibitor) (Experimental): CONDITIONING REGIMEN: Patients receive fludarabine phosphate IV on days -7 to -3, busulfan IV on days -6 to -3, and bortezomib IV on day -2.
  GVHD PROPHYLAXIS: Patients receive thymoglobulin IV on days -3 to -1, sirolimus PO on day -3, and tacrolimus IV on day -3. Patients undergo allogeneic HSCT on day 0.
  Interventions: Other: pharmacological study; Drug: tacrolimus; Drug: sirolimus; Biological: anti-thymocyte globulin; Drug: fludarabine phosphate; Drug: busulfan; Drug: bortezomib; Procedure: allogeneic hematopoietic stem cell transplantation; Other: laboratory biomarker analysis

INTERVENTIONS:
Other: pharmacological study — Correlative studies
  Other Names: pharmacological studies
Drug: tacrolimus — Given IV
  Other Names: FK 506; Prograf
Drug: sirolimus — Given PO
  Other Names: AY 22989; Rapamune; rapamycin; SLM
Biological: anti-thymocyte globulin — Given IV
  Other Names: ATG; ATGAM; lymphocyte immune globulin; Thymoglobulin
Drug: fludarabine phosphate — Given IV
  Other Names: 2-F-ara-AMP; Beneflur; Fludara
Drug: busulfan — Given IV
  Other Names: BSF; BU; Misulfan; Mitosan; Myeloleukon
Drug: bortezomib — Given IV
  Other Names: LDP 341; MLN341; VELCADE
Procedure: allogeneic hematopoietic stem cell transplantation — Undergo allogeneic HSCT
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
This pilot phase II trial studies how well giving high dose busulfan together with bortezomib works in treating patients with high risk multiple myeloma undergoing stem cell transplant. Drugs used in chemotherapy, such as busulfan, work in different ways to stop the growth of cancer cells, either by killing the cells or by stopping them from dividing. Bortezomib may stop the growth of cancer cells by blocking some of the enzymes needed for cells growth. Giving busulfan together with bortezomib before a stem cell transplant may kill more cancer cells

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine time to engraftment absolute neutrophil count (> 0.5 x 10^9/L for 3 consecutive days), and platelet (> 20X 109^/L for 3 consecutive days).

2. Incidence and severity of acute graft-versus-host disease (GVHD) using fludarabine (fludarabine phosphate) / busulfan / bortezomib preparative regimen and triple immune suppression with tacrolimus, sirolimus and Thymoglobulin (anti-thymocyte globulin).

3. To determine the safety related to this combination in the first six months post transplant, specifically, treatment related mortality and grade III and IV non hematologic toxicities, based on Common Terminology Criteria for Adverse Events (CTCAE) version 4 (v4).

SECONDARY OBJECTIVES:

I. Incidence of myeloma progression in this high risk group of patients.

II. Incidence of transplant related mortality and morbidity.

III. Incidence of thrombotic thrombocytopenic purpura (TTP) and sinusoidal obstructive syndrome (SOS).

IV. Incidence and severity of chronic GVHD.

V. Incidence of opportunistic infections including cytomegalovirus (CMV), herpes simplex virus (HSV), and Epstein-Barr virus (EBV) reactivation.

I. Overall and progression free survival (PFS) at Day 100, 6 months, 1 & 2 years post transplant.

VII. To determine recovery of T-cell, B cell, and natural killer (NK) cell phenotypes post transplant.

OUTLINE:

CONDITIONING REGIMEN: Patients receive fludarabine phosphate intravenously (IV) on days -7 to -3, busulfan IV on days -6 to -3, and bortezomib IV on day -2.

GVHD PROPHYLAXIS: Patients receive anti-thymocyte globulin IV on days -3 to -1, sirolimus orally (PO) on day -3, and tacrolimus IV on day -3. Patients undergo allogeneic hematopoietic stem cell transplantation (HSCT) on day 0.

After completion of study treatment, patients are followed up for up to 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Ability to provide informed consent
* Karnofsky Performance Status (KPS) >= 70
* Eastern Cooperative Oncology Group (ECOG) performance status =< 2
* Availability of a suitable allogeneic hematopoietic stem cell donor; minimum of human leukocyte antigen (HLA) 7/8 matched related or unrelated donor
* High risk multiple myeloma with poor prognostic features based on having one or more of the following criteria:
* Progressive disease after autologous transplant. No less than 3 months post auto transplant
* Progressive or stable disease after induction chemotherapy using the most potent myeloma agents Lenalidomide and/or Bortezomib
* Patients with high risk cytogenetic abnormalities documented on conventional cytogenetics or fluorescence in situ hybridization (FISH) (hypodiploidy, t(4:14), t(14:16) chromosome translocation, p53 and or complex cytogenetics) additionally, chromosome 13 deletion by standard cytogenetics
* Negative beta-human chorionic gonadotropin (β-HCG) pregnancy test for women, as well as implementation of birth control for men and women

Exclusion Criteria:

* Patients with prior allogeneic transplant, or more than one prior autologous transplant for any medical reason
* Prior treatment with busulfan or gemtuzumab (Mylotarg ®) for any reason
* Patient with history of allergy to boron, mannitol, or bortezomib
* Creatinine clearance (CrCl) =< 50 ml/min
* Ejection Fraction < 50%
* Diffusion capacity of carbon monoxide (DLCO) < 50% predicted
* Forced expiratory volume in 1 second (FEV1) < 50% predicted
* Forced vital capacity (FVC) < 50% predicted
* Patients with uncontrolled arrhythmia or uncontrolled heart disease at the screening time; patients with coronary heart disease (recent myocardial infarctions, angina, cardiac stent, or bypass surgery in the last 6 months) need to be cleared with a stress echo or nuclear myocardial perfusion stress test, and cardiology consult; all other cardiac history will be at the discretion of the principal investigator
* Liver enzymes > 3 times upper limit normal
* Bilirubin > 2 mg/dl (except Gilbert's disease)
* International normalized ratio (INR) > 2
* Any previous history of liver failure, hepatitis, or cirrhosis
* Systemic Amyloidosis Known history of hepatitis B, C, human immunodeficiency virus (HIV) or any current uncontrolled infection
* Grade > I neuropathy
* Women who are pregnant or lactating
* Current or history of alcohol or drug abuse
* Use of other investigational agents within 30 days of enrollment to this study
* Any patient with ascites
* Any patient on home oxygen
* Any clinical findings on history or physical exam which would in the opinion of the treating physician or principal investigator preclude the patient from participating in the study

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2012-02; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Zaid Al-Kadhimi, Principal Investigator — Barbara Ann Karmanos Cancer Institute
Locations (1):
- Barbara Ann Karmanos Cancer Institute, Detroit, Michigan, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Cancer center clinic.
Groups:
- Treatment (Chemotherapy, Enzyme Inhibitor): CONDITIONING REGIMEN: Patients receive fludarabine phosphate IV on days -7 to -3, busulfan IV on days -6 to -3, and bortezomib IV on day -2.
  GVHD PROPHYLAXIS: Patients receive thymoglobulin IV on days -3 to -1, sirolimus PO on day -3, and tacrolimus IV on day -3. Patients undergo allogeneic HSCT on day 0.
  anti-thymocyte globulin : Given IV
  pharmacological study : Correlative studies
  fludarabine phosphate : Given IV
  busulfan : Given IV
  bortezomib : Given IV
  allogeneic hematopoietic stem cell transplantation : Undergo allogeneic HSCT
  tacrolimus : Given IV
  laboratory biomarker analysis : Correlative studies
  sirolimus : Given PO
Period: Overall Study
Arm/Group | Treatment (Chemotherapy, Enzyme Inhibitor)
Started | 1
Completed | 1
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Chemotherapy, Enzyme Inhibitor)
Number analyzed (Participants) | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 46 (0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 1
Region of Enrollment [Number; unit: participants]
  United States | 1

OUTCOME MEASURES:

1. Primary Outcome: Incidence and Severity of Acute GVHD Using Fludarabine Phosphate / Busulfan / Bortezomib Preparative Regimen and Triple Immune Suppression With Tacrolimus, Sirolimus and Anti-thymocyte Globulin
Description: Graded using the Glucksberg scale. Proportions and confidence intervals will be estimated. Estimated using binary proportion estimates as well as competing risk method.
Time Frame: First 6 months post-transplant
Population: Data was not collected, because funding was unavailable to continue study.
Arm/Group | Treatment (Chemotherapy, Enzyme Inhibitor)
Number analyzed (Participants) | 0

2. Primary Outcome: Time to Platelet Absolute Neutrophil Recovery (Engraftment)
Description: Estimated using Kaplan-Meier method.
Time Frame: First 6 months post-transplant
Arm/Group | Treatment (Chemotherapy, Enzyme Inhibitor)
Number analyzed (Participants) | 0

3. Primary Outcome: Treatment Related Mortality Defined as Death in Continuous or Complete Remission
Description: Based on National Cancer Institute (NCI) CTCAE version 4.
Time Frame: From the date of transplant to the date of death, assessed up to 6 months post transplant
Arm/Group | Treatment (Chemotherapy, Enzyme Inhibitor)
Number analyzed (Participants) | 0

4. Primary Outcome: Grade III and IV Non Hematologic Toxicities
Description: Based on NCI CTCAE version 4.
Time Frame: First 6 months post transplant
Arm/Group | Treatment (Chemotherapy, Enzyme Inhibitor)
Number analyzed (Participants) | 0

5. Secondary Outcome: Incidence of Myeloma Progression
Time Frame: Time to the first observation of disease progression/relapse post transplant, assessed up to 2 years post transplant
Arm/Group | Treatment (Chemotherapy, Enzyme Inhibitor)
Number analyzed (Participants) | 0

6. Secondary Outcome: Incidence of Transplant Related Mortality and Morbidity
Time Frame: Up to 2 years post transplant
Arm/Group | Treatment (Chemotherapy, Enzyme Inhibitor)
Number analyzed (Participants) | 0

7. Secondary Outcome: Incidence of TTP
Time Frame: Up to 2 years post transplant
Arm/Group | Treatment (Chemotherapy, Enzyme Inhibitor)
Number analyzed (Participants) | 0

8. Secondary Outcome: Incidence of SOS
Time Frame: Up to 2 years post transplant
Arm/Group | Treatment (Chemotherapy, Enzyme Inhibitor)
Number analyzed (Participants) | 0

9. Secondary Outcome: Incidence and Severity of Chronic GVHD
Time Frame: Up to 2 years post transplant
Arm/Group | Treatment (Chemotherapy, Enzyme Inhibitor)
Number analyzed (Participants) | 0

10. Secondary Outcome: Incidence of Opportunistic Infections Including CMV, HSV, and EBV Reactivation
Time Frame: Weekly to day 100
Arm/Group | Treatment (Chemotherapy, Enzyme Inhibitor)
Number analyzed (Participants) | 0

11. Secondary Outcome: Overall Survival
Time Frame: Up to 2 years post transplant
Arm/Group | Treatment (Chemotherapy, Enzyme Inhibitor)
Number analyzed (Participants) | 0

12. Secondary Outcome: Progression Free Survival
Time Frame: From the day of transplant to progression, death, or last contact, assessed up to 2 years
Arm/Group | Treatment (Chemotherapy, Enzyme Inhibitor)
Number analyzed (Participants) | 0

13. Secondary Outcome: Recovery of T-cell, B Cell and NK Cell Phenotypes
Time Frame: Days 30, 60, 90, and at 6 months after transplant
Arm/Group | Treatment (Chemotherapy, Enzyme Inhibitor)
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Arm/Group | Treatment (Chemotherapy, Enzyme Inhibitor)
Serious Adverse Events (participants affected / at risk) | 1/1
Other Adverse Events (participants affected / at risk) | 0/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Chemotherapy, Enzyme Inhibitor) (N=1)
Mucositis oral (Gastrointestinal disorders) | 1 (1)
Fever (General disorders) | 1 (2)
Staphylococcus bacteremia (Infections and infestations) | 1 (1)
CMV (Infections and infestations) | 1 (1)
Headache (Nervous system disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
Data was not collected, because funding was unavailable to continue study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes